CLINICAL TRIAL: NCT05389189
Title: A Tailored Psychological Intervention (MITIG.RA) for Managing Fatigue in Rheumatoid Arthritis: Protocol for a Randomized Controlled Trial
Brief Title: A Tailored Psychological Intervention (MITIG.RA) for Managing Fatigue in Rheumatoid Arthritis
Acronym: CoMIRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, José António Pereira da Silva, Professor, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBS.SF.01/2021
Record Dates: First submitted 2022-03-24; First posted 2022-05-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Contextual-cognitive behavioural; Fatigue
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Care (Active Comparator): Intervention content
  The MITIG.RA program incorporates the following key topics during the 8 weeks of intervention (1st phase):
  (i) Psychoeducation on RA, sleep hygiene, exercise, and general nutritional recommendations (promote behavioural change and self-care, boost the sense of self-worth and self-efficacy) (ii) Activity engagement and pacing (iii) The functioning of the mind and its problematic patterns (iv) Focusing on the 'here and now' (mindfulness) (v) Learning new ways of self-relating - self-compassion (vi) Making room for suffering (acceptance); and (vii) Moving towards what matters (identification of valued life directions and promotion of consistent values and goals-directed behaviour).
  Booster sessions, at 4 and 12 weeks after completion of the first phase
  Interventions: Behavioral: Intervention Arm
- TAU Care (No Intervention): Usual Care respecting international recommendations for the management of RA.

INTERVENTIONS:
Behavioral: Intervention Arm — The MITIG.RA program incorporates the following key topics during the 8 weeks of intervention (1st phase):
  (i) Psychoeducation on RA, sleep hygiene, exercise, and general nutritional recommendations (promote behavioural change and self-care, boost the sense of self-worth and self-efficacy) (ii) Activity engagement and pacing (iii) The functioning of the mind and its problematic patterns (iv) Focusing on the 'here and now' (mindfulness) (v) Learning new ways of self-relating - self-compassion (vi) Making room for suffering (acceptance); and (vii) Moving towards what matters (identification of valued life directions and promotion of consistent values and goals-directed behaviour).
  Arms: CBT Care

SUMMARY:
The objective of this study is to examine the efficacy of the Compassion and Mindfulness Intervention for RA (MITIG.RA), a novel intervention combining different components of Cognitive Behavioural Therapy (CBT), compared to treatment-as-usual (TAU) in the management of Rheumatoid Arthritis (RA) associated fatigue.

This is a multicentre, two-arm parallel randomized controlled trial. Patients will be screened for eligibility, willingness to participate, and will be assessed and randomized to the experimental (MITIG.RA + TAU) or control condition (TAU) using computer-randomization. MITIG.RA will be delivered by a certified psychologist and comprises eight sessions of 2 hours, followed by two booster sessions. Outcomes will be assessed via validated self-report measures and include levels of fatigue (primary outcome), perceived impact of disease, depressive symptoms, mindfulness, self-compassion, safety, and satisfaction (secondary outcomes). Assessment will take place at baseline, post-intervention, before the first and second booster session (week 12 and 20, respectively), and at 32 and 44 weeks after the interventions' beginning.

DETAILED DESCRIPTION:
Primary aim: to investigate the impact of the program Compassion and Mindfulness Intervention for RA (MITIG.RA) in RA-associated fatigue in comparison to treatment as usual (TAU).

Secondary aims: the effects the intervention has upon the patient's satisfaction with disease status, overall perceived impact of disease, depression and anxiety levels, and self-compassion skills.

Methods Selection of patients: Adult patients with RA, currently in PGA-near-remission; Rheumatoid Arthritis Impact of disease (RAID) - fatigue ≥ 3; Patient Experienced Symptom State (PESS) < "good" and under stable medication (at least 3 months).

Study design: two-arm parallel superiority randomized controlled trial. Participants will be randomized (1:1) into one of two conditions: the experimental condition (CoMIRA Program plus TAU]) and the control condition (TAU only).

Intervention: delivered in a group sessions, online, for eight consecutive weeks, followed by two booster sessions after 4 and 12 additional weeks.

Active Group: The MITIG.RA program incorporates the following key topics during the 8 weeks of intervention (1st phase):

(i) Psychoeducation on RA, sleep hygiene, exercise, and general nutritional recommendations (promote behavioural change and self-care, boost the sense of self-worth and self-efficacy) (ii) Activity engagement and pacing (iii) The functioning of the mind and its problematic patterns (iv) Focusing on the 'here and now' (mindfulness) (v) Learning new ways of self-relating - self-compassion (vi) Making room for suffering (acceptance); and (vii) Moving towards what matters (identification of valued life directions and promotion of consistent values and goals-directed behaviour).

The closing session comprises a review of the main concepts and "take-home" messages, discussion of potential setbacks and strategies to deal with them, and participant's feedback on the intervention and the progress made.

The booster sessions, at 4 and 12 weeks after completion of the first phase, will focus on the revision of previously learned concepts, evaluation of potential barriers/difficulties encountered, strategies employed to deal with them, and clarification of any impending question.

Comparison: Usual Care

Procedure: The participants who accept to participate will be randomized (1:1). sessions will be delivered via zoom, in a group format. Patients will be assessed at baseline, post-intervention, before the first and second booster session (week 12 and 20, respectively), and at 32 and 44 weeks after the interventions' beginning.

Analysis: An intention-to-treat analysis will be conducted whenever possible and complemented with per-protocol analysis if needed. Analysis of covariance (ANCOVA) will be used to assess between-group differences in fatigue scores (the primary outcome) at 3-month follow-up after the second booster session (32nd week), controlling for baseline values. The same analytic procedure will be used to examine between-group differences in perceived disease activity, depression, mindfulness, and self-compassion (secondary outcomes) at the 32nd week. All effect sizes will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the 1987 ACR or 2010 ACR/EULAR classification criteria for RA;
* In PGA-near remission: Tender and swollen 28 joint counts and C-reactive protein (CRP) (mg/dl) < 1, and Patient Global Assessment of disease Activity (PGA > 1,
* RAID - fatigue ≥ 3;
* PESS < "good"
* Under stable medication (at least 3 months).

Exclusion Criteria:

* Less than 6 years of formal education;
* Unable to attend zoom meetings unaided;
* Unable to fulfil self-report questionnaires unaided;
* Pain-related comorbidities (e.g. fibromyalgia or osteoarthritis)
* Presence of other comorbid medical conditions that may cause fatigue, such as anaemia (Hb<10mg/dL), uncontrolled hypothyroidism or cancer;
* Presence of severe psychological symptoms or disorders (e.g. psychosis, severe depression, substance abuse);
* Currently ongoing psychological interventions or formal psychiatric treatment;
* Pregnant patients;
* Otherwise disabled patients (advanced articular/bone erosion);
* Refuse to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Week 32
  Fatigue levels will be assessed by the 0-10 numerical rating scale assessing fatigue as part of the RAID.7.Higher Scores indicate higher levels of fatigue

SECONDARY OUTCOMES:
Satisfaction With Disease Status- PESS | Week 32
  The Patient Experienced Symptom State (PESS), evaluates the degree of satisfaction of the patients with the status of RA during the last week, through a single item rated on a 5-level Likert scale response ('very bad', 'bad', 'acceptable', 'good' and 'very good').
Perceived Impact of the Disease | Week 32
  Assessed through the Rheumatoid Arthritis Impact of Disease (RAID) score and its individual domains (RAID.7). The RAID is a 7-item patient-derived measure designed to evaluate the perceived impact of RA upon important health-related domains, namely pain, functional disability, fatigue, sleep, physical well-being, emotional well-being, and coping. The items are rated using 11-points numeric rating scales (0 to 10). Domains can be combined into a single score (RAID) or used separately (RAID.7). Higher scores indicate greater impact of disease.
Anxiety and Depression Levels | Week 32
  Assessed through the Hospital Anxiety Depression Scale (HADS). This scale comprises 14 items, rated on a 4-point Likert scale, aimed at screening for the presence and severity of anxiety and depressive symptoms in the last 7 days. The score range between 0-21 for each condition, with higher values are indicative of more severe levels of symptoms, with a cut-off score of 11 being indicative of a probable diagnosis of depressive major episode.
Self-Compassion | Week 32
  Self-compassion will be assessed by the Self-Compassion Scale (SCS). This 12-item measure is a shorter form of the original scale developed and aims to assess the type of relationship one establishes with oneself in the face of setbacks or difficult times. Items are rated on a 5-point Likert scale. Total score is calculated through the average of the 12 items, ranging from 1 to 5, with greater values indicating greater levels of self-compassion.
Affective Mindfulness | Week 32
  Active Mindfulness will be assessed through the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT) is a 23-itens self-report measure aimed at assessing psychological flexibility. Items are rated using a 7-point response scale from 0 ('Strongly disagree') to 7 ('Strongly agree'). The scale comprises 3 factors, namely: openness to experience, behavioral awareness and valued action. Scores range from 0-60 (openness to experience subscale), 0-30 (behavioral awareness subscale), 0-48 (valued action subscale), and 0-138 (total score), and are computed by summing all respective items. Higher scores indicate greater psychological flexibility.
Adverse Events | Week 32
  Safety-related outcomes will be evaluated through participants' reporting of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jose AP daSilva, PhD, Principal Investigator — CHUC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duarte C, Spilker RLF, Paiva C, Ferreira RJO, da Silva JAP, Pinto AM. MITIG.RA: study protocol of a tailored psychological intervention for managing fatigue in rheumatoid arthritis randomized controlled trial. Trials. 2023 Oct 6;24(1):651. doi: 10.1186/s13063-023-07692-4. PMID 37803467